CLINICAL TRIAL: NCT03999190
Title: Imaging Dopamine D2 Agonist Binding Sites in Schizophrenia
Status: Withdrawn | Type: Observational
Why Stopped: investigational radiotracer was not approved
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 18-01207
Record Dates: First submitted 2019-06-11; First posted 2019-06-26 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Dextroamphetamine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 30 subjects with schizophrenia
  Interventions: Drug: NPA radiotracer; Drug: Raclopride radiotracer; Drug: Dextroamphetamine
- 30 healthy controls
  Interventions: Drug: NPA radiotracer; Drug: Raclopride radiotracer; Drug: Dextroamphetamine

INTERVENTIONS:
Drug: NPA radiotracer — [11C]NPA radiotracer, 2 injection per subject
  Antagonist ([11C]raclopride) and agonist ([11C]NPA) radiotracer will be used sequentially to measure binding potential (BPND) under baseline conditions and 3-hours following oral administration of 0.5 mg/kg amphetamine in the same 30 medication free subjects with schizophrenia (MF-S) and 30 healthy control subjects (HC).
Drug: Raclopride radiotracer — [11C]raclopride radiotracer, 2 injections per subject
  Antagonist ([11C]raclopride) and agonist ([11C]NPA) radiotracer will be used sequentially to measure binding potential (BPND) under baseline conditions and 3-hours following oral administration of 0.5 mg/kg amphetamine in the same 30 medication free subjects with schizophrenia (MF-S) and 30 healthy control subjects (HC).
Drug: Dextroamphetamine — Dextroamphetamine, one oral administration of 0.5 mg/kg per subject Antagonist ([11C]raclopride) and agonist ([11C]NPA) radiotracer will be used sequentially to measure binding potential (BPND) under baseline conditions and 3-hours following oral administration of 0.5 mg/kg amphetamine in the same 30 medication free subjects with schizophrenia (MF-S) and 30 healthy control subjects (HC).

SUMMARY:
The goals of this study is to determine (1) if differences in D2/3 receptor affinity states exist between medication-free subjects with SCH (MF-S) compared with healthy controls (HC), (2) the degree to which pre- and post-synaptic factors contribute to increased striatal dopamine (DA) signaling in MF-S and (3) to test the hypotheses that optimal DA transmission in the dorsal caudate (DCA) is necessary for normal working memory (WM) function.

DETAILED DESCRIPTION:
An antagonist ([11C]raclopride) and agonist ([11C]NPA) radiotracer will be used sequentially, in a counterbalanced design, to measure binding potential (BPND) under baseline conditions and 3-hours following oral administration of 0.5 mg/kg amphetamine in the same 30 MF-S and 30 HC. The main outcome measures will be baseline BPND and the percent change in BPND induced by amphetamine, denoted ∆BPND, in the subdivisions of the striatum. In addition, all subjects will undergo fMRI while performing a WM task concurrent with both the initial pre- and initial post-amphetamine PET scans to explore the relationship between DCA DA transmission and fMRI BOLD response in the dorsal lateral prefrontal cortex (DLPFC) during a WM task.

ELIGIBILITY:
Inclusion Criteria:

* HEALTHY CONTROLS

  1. Males or females between 18 and 35 years old (History)
  2. Absence of current (i.e. last six months) psychiatric conditions (including alcohol and drug abuse). Subjects with a history of a non-psychotic psychiatric disorder who have been asymptomatic and not taking medication for the past 6 months may be eligible.

     (History, SCID-NP (non-patient version))
  3. A negative urine toxicology with the exception of cannabis; in the case of a positive urine cannabis test a salivary cannabis test will be administered on the day of the PET scans to ensure subjects have not used within 24 - 48 hours.

     (Urine toxicology)
  4. Medically Healthy (History, EKG, physical, labs (detailed labs are listed under screening procedures))
  5. Weight between 44 and 115 kg (physical exam)
  6. Baseline systolic BP of < 150 and > 100, diastolic BP < 90 and >60 and baseline HR less than 90 (Physical exam)
* SUBJECTS WITH SCHIZOPHRENIA Criteria (Assessment)

  1. Males or females between 18 and 35 years old (History)
  2. Fulfill DSM-V criteria for schizophrenic illness, schizophreniform or schizoaffective disorder (History, SCID)
  3. A negative urine toxicology with the exception of cannabis; in the case of a positive urine cannabis test a salivary cannabis test will be administered on the day of the PET scans to ensure subjects have not used within 24 - 48 hours.

     (Urine toxicology)
  4. Medically Healthy (History, EKG, physical, labs (detailed labs are listed in screening procedures))
  5. Clinical Global Impression-Severity scale (CGI-S) less than or equal to 4 (moderately ill).
  6. Off all medications for at least 1 week, does not wish to restart medications immediately and clinically stable while off medications. With the exception of lorazepam at a maximal dose of 2 mg QD, up to 24 h prior to the scans, and absence of injection of depot medication within the last 6 months (Interview and discussion with treating clinician)
  7. Weight between 44 and 115 kg (Physical exam)
  8. Baseline systolic BP of < 150 and > 100, diastolic BP < 90 and >60 and baseline HR less than 90 (Physical exam)

Exclusion Criteria:

* HEALTHY CONTROLS

  1. Pregnancy or lactation, lack of effective birth control during 15 days before the scans* (Blood or Urine pregnancy test, history)
  2. Presence or positive history of serious medical or neurological illness, including low hemoglobin and seizure history.

     (Medical and neurological history, EKG, blood tests)
  3. Any current use (within past month) of amphetamines, opiates, cocaine, sedative-hypnotics, ecstasy PCP.

     (History, urine toxicology)
  4. Any use of cannabis beyond occasional use (i.e. more than 2 - 4 times per month) (History, saliva cannabis test)
  5. Metal implants or paramagnetic objects contained within the body which may interfere with the MRI scan (but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant. Dental fillings do not present a risk for MRI), as determined in consultation with a neuroradiologist and according to the guidelines set forth in the following reference book commonly used by neuroradiologists: "Guide to MR procedures and metallic objects" Shellock, PhD, Lippincott Williams and Wilkins, NY 2001. If there is any doubt, subjects will be excluded.

     (Interview and history)
  6. Lifetime exposure to radiation in the workplace; or participation in research protocols involving exposure to radiation within the previous year such that the total cumulative annual radiation dose (i.e., from participation in the previous research studies and this study) would exceed the radiation dose limits specified in the FDA regulations at 21 CFR 361.1, Radioactive Drugs Considered Generally Safe and Effective (i.e. annual cumulative radiation dose limit = 5 rems to gonads, blood-forming organs, lens of eye, whole body; 15 rems to other organs).

     (Interview and history)
  7. Medical history of chronic obstructive pulmonary disease or other chronic respiratory disorders (Medical history)
  8. More than one risk factor for coronary artery disease (smoking, cholesterol > 240 mg/dl, sedentary lifestyle) baseline SBP > 140 of DBP> 90) (History, physical examination and blood chemistry)
  9. Positive Allen Test indicating lack of collateral flow to hand (Physical Exam)
  10. Subjects with family history of a psychotic disorder, drug and alcohol Abuse/Dependence in first-degree relatives. (History)
* SUBJECTS WITH SCHIZOPHRENIA Criteria (Assessment)

  1. DSM-V disorder other than schizophrenia, schizophreniform or schizoaffective disorder (History, SCID)
  2. Any current use (within past month) of amphetamines, opiates, cocaine, sedative-hypnotics, ecstasy PCP.

     (History, urine toxicology)
  3. Any use of cannabis beyond occasional use (i.e. more than 2 - 4 times per month) (History, saliva cannabis test)
  4. Antipsychotic medications in the last 3 weeks (6 months for depot medications) prior to the first PET scanning session.

     (History)
  5. Pregnancy or lactation, lack of effective birth control - OCP are allowed. (Pregnancy test, history)
  6. Presence or positive history of severe medical or neurological illness or any cardiovascular disease, low hemoglobin, and seizure history.

     (Medical and neurological history, neurological exam, EKG, blood chemistry)
  7. Lack of capacity to give informed consent (Interview)
  8. History of significant violent or suicidal behavior (Interview and review of records)
  9. Metal implants or paramagnetic objects contained within the body which may interfere with the MRI scan (but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant. Dental fillings do not present a risk for MRI), as determined in consultation with a neuroradiologist and according to the guidelines set forth in the following reference book commonly used by neuroradiologists: "Guide to MR procedures and metallic objects" Shellock, PhD, Lippincott Williams and Wilkins, NY 2001. If there is any doubt, subjects will be excluded.

     (Interview and history)
  10. Lifetime exposure to radiation in the workplace; or participation in research protocols involving exposure to radiation within the previous year such that the total cumulative annual radiation dose (i.e., from participation in the previous research studies and this study) would exceed the radiation dose limits specified in the FDA regulations at 21 CFR 361.1, Radioactive Drugs Considered Generally Safe and Effective (i.e. annual cumulative radiation dose limit = 5 rems to gonads, blood-forming organs, lens of eye, whole body; 15 rems to other organs).

      (Interview and history)
  11. Medical history of chronic obstructive pulmonary disease or other chronic respiratory disorders (Medical history)
  12. More than one risk factor for coronary artery disease (smoking, cholesterol > 240 mg/dl, sedentary lifestyle) baseline SBP > 140 of DBP> 90) (History, physical examination and blood chemistry)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: SCHIZOPHRENIA patiens 18-35; Healthy Controls 18-35
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
base line Binding Potential (BPND) | 37 Days
  PET outcome measure of the density of "available" neuroreceptors and the affinity of a drug to that neuroreceptor.
percent change in BPND | 37 Days
  Difference between BPND measured in the post-amphetamine condition (BPND AMPH) and BPND measured in the baseline condition (BPND BASE) expressed as a percentage of BPND BASE: BPND = 100 * (BPND AMPH - BPND BASE)/BPND BASE.

CONTACTS AND LOCATIONS:
Overall Officials: William Frankle, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States